CLINICAL TRIAL: NCT02716142
Title: Rectal Misoprostol Versus Sublingual Misoprostol in Decreasing Blood Loss Prior to Abdominal Myomectomy: A Randomized Double-blinded Clinical Trial
Brief Title: Rectal Misoprostol Versus Sublingual Misoprostol Prior to Myomectomy
Acronym: RM-SLM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MISOP
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Bleeding During Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): rectal misoprostol 400 microgram
  Interventions: Drug: rectal misoprostol
- Group B (Active Comparator): sublingual misoprostol 400 microgram
  Interventions: Drug: sublingual misoprostol

INTERVENTIONS:
Drug: rectal misoprostol — patients will take 2 tablets of rectally misoprostol 400 microgram 60 minutes before the procedure
  Arms: Group A
Drug: sublingual misoprostol — patients will take 2 tablets of sublingual misoprostol 400 microgram 60 minutes before the procedure
  Arms: Group B

SUMMARY:
the aim of the study is To compare the effectiveness of rectally administered prostaglandin E1 synthetic analogue (misoprostol) 400 microgram versus sublingually administered misoprostol before myomectomy to decrease blood loss during and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging
* Age ≥ 18 years and ≤ 50 years
* Pre-operative hemoglobin >8 g/dl
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history
* Five or less symptomatic uterine myomas
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks pregnancy

Exclusion Criteria:

* Patients who have had a prior abdominal myomectomy
* Post-menopausal women
* Patients with known bleeding/clotting disorders
* Patients with a history of gynecologic malignancy
* Hypertension.
* Cardiac and Pulmonary diseases.
* Obesity (body mass index > 30 kg/m2).
* History of allergic reactions attributed to misoprostol
* Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Mean amount of blood loss | intraoperative

SECONDARY OUTCOMES:
Change of hemoglobin level | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided